CLINICAL TRIAL: NCT04002401
Title: A Phase 2 Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Axicabtagene Ciloleucel in Combination With Rituximab in Participants With Refractory Large B-Cell Lymphoma (ZUMA-14)
Brief Title: Safety and Efficacy of Axicabtagene Ciloleucel in Combination With Rituximab in Participants With Refractory Large B-Cell Lymphoma
Acronym: ZUMA-14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-471-0114; 2019-004803-11 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Refractory Large B-cell Lymphoma
MeSH Terms: interventions — axicabtagene ciloleucel; Rituximab; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleucel and Rituximab Combination (Experimental): Participants will receive rituximab 375 mg/m^2, once on Day -5 along with conditioning chemotherapy (fludarabine 30 mg/m^2 over 30 minutes and cyclophosphamide 500 mg/m^2 over 60 minutes) once on Days -5 to -3, followed by axicabtagene ciloleucel 2 x 10^6 anti-cluster of differentiate 19 (CD19) chimeric antigen receptor (CAR) T cells/kg once on Day 0 and additional rituximab 375 mg/m^2 of 5 doses, once every 28 days starting from Day 21 up to Day 133.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Rituximab; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — A single infusion of CAR-transduced autologous T cells administered intravenously
  Other Names: Yescarta®
Drug: Rituximab — Administered intravenously
  Other Names: RITUXAN®
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
The primary objective of this study is to estimate the efficacy of axicabtagene ciloleucel in combination with rituximab, as measured by assessment of response rates in adult participants with relapsed/refractory large B-cell lymphoma.

DETAILED DESCRIPTION:
Following at least 24 months of assessments after axicabtagene ciloleucel infusion, participants will be asked to rollover to a separate long-term follow-up study (Study KT-US-982-5968). Participants will complete the remainder of the 15-year follow-up assessments in the KT-US-982-5968 study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed large B-cell lymphoma
* Chemotherapy-refractory disease, defined as one or more of the following:

  * No response to first-line therapy (primary refractory disease)
  * No response to second or greater lines of therapy OR
  * Refractory after autologous stem cell transplant (ASCT)
* At least 1 measureable lesion according to the Lugano Classification (Cheson 2014).
* Individuals must have received adequate prior therapy, including at a minimum:

  * Anti-CD20 monoclonal antibody
  * An anthracycline-containing chemotherapy regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate renal, hepatic, pulmonary, and cardiac function

Key Exclusion Criteria:

* Known CD19 negative or CD20 negative tumor
* History of Richter's transformation of Chronic Lymphocytic Leukemia (CLL)
* Prior CAR therapy or other genetically modified T-cell therapy
* Prior organ transplantation including prior allogeneic stem cell transplant (SCT)
* Prior CD19 targeted therapy
* Clinically significant infection or cardiopulmonary disease
* Presence of any in-dwelling lines or drains (dedicated central venous access catheters allowed)
* History or presence of central nervous system (CNS) lymphoma or nonmalignant CNS disorder or cerebrospinal fluid (CSF) malignant cells or brain metastases
* History of autoimmune disease
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the last 6 months

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (14):
- United States (14):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York Presbyterian Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Strati P, Leslie L, Shiraz P, Budde LE, Oluwole OO, Ulrickson M, Ramakrishnan A, Zhang T, Sun J, Milletti F, Kanska J, Shen R, Neumann F, Xu H, Patel K. Axicabtagene ciloleucel in combination with rituximab for refractory large B cell lymphoma: the phase 2, single-arm ZUMA-14 trial. Nat Cancer. 2026 Jan 5. doi: 10.1038/s43018-025-01102-1. Online ahead of print. PMID 41492094
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-471-0114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 36 participants were screened.
Groups:
- Axicabtagene Ciloleucel and Rituximab Combination: Participants received rituximab 375 mg/m^2 intravenously (IV) once on Day -5 along with conditioning chemotherapy (fludarabine 30 mg/m^2 over 30 minutes and cyclophosphamide 500 mg/m^2 over 60 minutes) administered IV once on Days -5 to -3, followed by axicabtagene ciloleucel 2 x 10^6 anti-cluster of differentiate 19 (CD19) chimeric antigen receptor (CAR) T cells/kg administered IV once on Day 0 and additional rituximab 375 mg/m^2 of 5 doses, administered IV once every 28 days starting from Day 21 up to Day 133.
Period: Overall Study
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Started | 27
Completed | 0
Not Completed | 27
Not completed — Rolled Over to Long-term Follow-up Study | 13
Not completed — Death | 10
Not completed — Subject Withdrawal of Consent From Further Follow-up | 2
Not completed — Enrolled but Never Treated | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants treated with any dose of axicabtagene ciloleucel.
Groups:
- Axicabtagene Ciloleucel and Rituximab Combination: Participants received rituximab 375 mg/m^2 IV once on Day -5 along with conditioning chemotherapy (fludarabine 30 mg/m^2 over 30 minutes and cyclophosphamide 500 mg/m^2 over 60 minutes) administered IV once on Days -5 to -3, followed by axicabtagene ciloleucel 2 x 10^6 anti-CD19 CAR T cells/kg administered IV once on Day 0 and additional rituximab 375 mg/m^2 of 5 doses, administered IV once every 28 days starting from Day 21 up to Day 133.
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19
  Race: Other or More Than One Race | 4
  Race: Asian | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate Per the International Working Group (IWG) Lugano Classification as Determined by Study Investigators
Description: CR rate is defined as the incidence of a CR per the IWG Lugano Classification as determined by study investigators. CR rate: percentage of participants with CR [complete metabolic response (CMR); complete radiological response (CRR)]. CMR: positron emission tomography (PET) 5-point scale (5-PS) scores of 1 (no uptake above background), 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass); no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow (BM). CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion (LDi); no extralymphatic sites of disease; absent non-measured lesion (NMLs); organ enlargement regress to normal; no new sites; and bone marrow normal by morphology. 95% confidence interval (CI) was calculated by Clopper-Pearson method.
Time Frame: First infusion date up to maximum duration of 32.7 months
Population: Modified intent-to-treat (mITT) analysis set included all enrolled participants who were treated with the target dose of axicabtagene ciloleucel and at least 1 dose of rituximab after axicabtagene ciloleucel infusion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
percentage of participants | 73 [52 to 88]

2. Secondary Outcome: Percentage of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant that does not necessarily have a relationship with study treatment or worsening of a pre-existing medical condition. TEAEs are any AEs with onset on or after axicabtagene ciloleucel infusion or worsening of a pre-existing medical condition that occurs on or after axicabtagene ciloleucel infusion.
Time Frame: First infusion date up to maximum duration of 27 months
Population: Safety analysis set included all participants treated with any dose of axicabtagene ciloleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Value
Description: Grading categories were determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Laboratory parameters with only non-zero values are presented.
Time Frame: First infusion date up to maximum duration of 27 months
Population: Participants in the safety analysis set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
percentage of participants
  Alanine Aminotransferase | 12
  Aspartate Aminotransferase | 12
  Bilirubin | 8
  Calcium | 8
  Direct Bilirubin | 15
  Glucose | 19
  Magnesium | 8
  Urate | 8

4. Secondary Outcome: Objective Response Rate (ORR) Per the IWG Lugano Classification as Determined by Study Investigators
Description: ORR: percentage of participants with CR [CMR;CRR] or PR [partial metabolic response (PMR); partial radiologic response (PRR)].CMR: PET 5PS scores of 1 (no uptake above background, 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass; no new lesions; no evidence of FDG-avid disease in BM. CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in LDi;no extralymphatic sites of disease;absent NMLs;organ enlargement regress to normal;no new sites;bone marrow morphology normal. PMR: scores 4 (uptake moderately > liver), 5 (uptake markedly > liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at end of treatment (EOT). PRR: ≥ 50% decrease in sum of the product of perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites; absent/normal, regressed, but no increase of NMLs; spleen regressed by > 50% in length beyond normal; no new sites.
Time Frame: First infusion date up to maximum duration of 32.7 months
Population: Participants in the mITT analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
percentage of participants | 88 [70 to 98]

5. Secondary Outcome: Duration of Response (DOR) Per the IWG Lugano Classification as Determined by Study Investigators
Description: DOR is defined only for participants who experience an objective response and is the time from the first objective response to disease progression [progressive metabolic disease (PMD); progressive radiologic disease (PRD)] or death from any cause. Objective response is defined in outcome measure (OM) 4. PMD: scores 4 (uptake moderately > liver), 5 (uptake markedly > liver, new lesions) with increased uptake compared with baseline; new fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma rather than another etiology; new or recurrent FDG-avid foci in bone marrow. PRD: LDi >1.5 cm; ≥ 50% increase from cross product of LDi and perpendicular diameter (PPD); increase in LDi or shortest axis perpendicular to the LDi (SDi) of 0.5 cm for lesions ≤1.5 cm and 1 cm for lesions >2 cm; spleen increased by >50% in length beyond normal; new or recurrent splenomegaly, bone marrow involvement; new lesions; progression of pre-existing lesions. Kaplan-Meier (KM) estimate of median was reported.
Time Frame: From the date of first confirmed objective response (CR or PR) to disease progression or death regardless of cause (up to approximately 32.7 months)
Population: Participants in the mITT analysis set with an objective response (CR+PR) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 23
months | 26.0 [2.6 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events.

6. Secondary Outcome: Progression-Free Survival (PFS) Per the IWG Lugano Classification as Determined by Study Investigators
Description: PFS is defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression (PMD; PRD) or death from any cause. PMD: scores 4 (uptake moderately > liver), 5 (uptake markedly > liver, new lesions) with increased uptake compared with baseline; new FDG-avid foci consistent with lymphoma rather than another etiology; new or recurrent FDG-avid foci in bone marrow. PRD: LDi >1.5 cm; ≥ 50% increase from cross product of LDi and PPD; increase in LDi or SDi of 0.5 cm for lesions ≤1.5 cm and 1 cm for lesions >2 cm; spleen increased by >50% in length beyond normal; new or recurrent splenomegaly, bone marrow involvement; new lesions; progression of pre-existing lesions. KM estimate of median was reported.
Time Frame: First infusion date up to disease progression or death regardless of cause (up to approximately 32.7 months)
Population: Participants in the mITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
months | 23.6 [3.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from axicabtagene ciloleucel infusion to the date of death from any cause. KM estimate of median was reported.
Time Frame: First infusion date up to death regardless of cause (up to approximately 32.7 months)
Population: Participants in the mITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
months | NA [25.8 to NA] — KM median and upper limit of 95% CI were not reached due to insufficient number of participants with events.

8. Secondary Outcome: Peak Level of Anti-CD19 CAR T Cells in Blood
Description: Peak was defined as the maximum number of CAR T cells in blood measured after infusion.
Time Frame: Baseline (Day 0), post-infusion on Days 7, 14, 21, 28, 49, 105, 180, Months 9, 12, 15, 18, and 24
Population: Participants in the safety analysis set were analyzed.
Measure: Median (Full Range); unit: cells per microliter (cells/µL)
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
cells per microliter (cells/µL) | 40.33 [1.15 to 304.36]

9. Secondary Outcome: Level of Anti-CD19 CAR T Cells in Blood by Visit
Time Frame: Baseline (Day 0), post-infusion on Days 7, 14, 21, 28, 49, 105, 180, Months 9, 12, 15, 18, and 24
Population: Participants in the safety analysis set with available data were analyzed.
Measure: Median (Full Range); unit: cells/µL
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
cells/µL
  Baseline (Day 0) | 0.00 [0.00 to 0.00]
  Day 7 Post-infusion: number analyzed (Participants) | 25
  Day 7 Post-infusion | 18.11 [1.15 to 304.36]
  Day 14 Post-infusion: number analyzed (Participants) | 20
  Day 14 Post-infusion | 12.74 [0.05 to 172.54]
  Day 21 Post-infusion: number analyzed (Participants) | 25
  Day 21 Post-infusion | 4.66 [0.02 to 43.26]
  Day 28 Post-infusion: number analyzed (Participants) | 25
  Day 28 Post-infusion | 1.66 [0.03 to 17.14]
  Day 49 Post-infusion: number analyzed (Participants) | 17
  Day 49 Post-infusion | 0.99 [0.01 to 26.49]
  Day 105 Post-infusion: number analyzed (Participants) | 19
  Day 105 Post-infusion | 0.32 [0.00 to 1.23]
  Day 180 Post-infusion: number analyzed (Participants) | 14
  Day 180 Post-infusion | 0.09 [0.00 to 1.34]
  Month 9 Post-infusion: number analyzed (Participants) | 14
  Month 9 Post-infusion | 0.06 [0.00 to 1.01]
  Month 12 Post-infusion: number analyzed (Participants) | 14
  Month 12 Post-infusion | 0.0054 [0.00 to 0.91]
  Month 15 Post-infusion: number analyzed (Participants) | 10
  Month 15 Post-infusion | 0.0027 [0.00 to 0.47]
  Month 18 Post-infusion: number analyzed (Participants) | 11
  Month 18 Post-infusion | 0.00 [0.00 to 0.36]
  Month 24 Post-infusion: number analyzed (Participants) | 9
  Month 24 Post-infusion | 0.00 [0.00 to 0.00]

10. Secondary Outcome: Area Under the Curve of CAR T Cells From Day 0 to Day 28 (AUC0-28)
Description: AUC0-28 is defined as the area under curve in a plot of number of CAR T cells against scheduled visit from Day 0 to Day 28.
Time Frame: Baseline (Day 0), post-infusion on Days 7, 14, 21, and 28
Population: Participants in the safety analysis set were analyzed.
Measure: Median (Full Range); unit: cells/μL*days
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
cells/μL*days | 376.83 [14.93 to 3430.50]

11. Secondary Outcome: Time to Peak Level of Anti-CD19 CAR T Cells in Blood
Description: Time to peak was defined as the number of days from the date of the axicabtagene ciloleucel infusion to the date of peak level defined as the maximum number of CAR T cells in blood measured after infusion.
Time Frame: Baseline (Day 0), post-infusion on Days 7, 14, 21, 28, 49, 105, 180, Months 9, 12, 15, 18, and 24
Population: Participants in the safety analysis set were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
Number analyzed (Participants) | 26
days | 8 [8 to 21]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Enrollment up to last follow up visit (maximum duration of 37.9 months); Adverse events: First infusion date up to maximum duration of 27 months
Description: All-cause mortality: All enrolled analysis set included all the enrolled participants.
  Adverse events: Safety analysis set included all participants treated with any dose of axicabtagene ciloleucel.
Arm/Group | Axicabtagene Ciloleucel and Rituximab Combination
All-Cause Mortality (participants affected / at risk) | 11/27
Serious Adverse Events (participants affected / at risk) | 14/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel and Rituximab Combination (N=26)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 3
Covid-19 pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Aphasia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel and Rituximab Combination (N=26)
Anaemia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 5
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Sinus tachycardia (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 8
Eye pain (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chills (General disorders) | 4
Fatigue (General disorders) | 10
Gait disturbance (General disorders) | 2
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 3
Pyrexia (General disorders) | 23
Hypogammaglobulinaemia (Immune system disorders) | 5
Covid-19 (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Aphasia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Encephalopathy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 6
Agitation (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT04002401/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04002401/SAP_001.pdf
  • Statistical Analysis Plan: Translational Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT04002401/SAP_002.pdf